CLINICAL TRIAL: NCT06683235
Title: Effect of Flaxseed Consumption as a Treatment for Adults With Type 2 Diabetes Mellitus in Oaxaca de Juárez, Oaxaca
Brief Title: Effect of Flaxseed as a Treatment for Adults With Type 2 Diabetes Mellitus in Mexico
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma Benito Juárez de Oaxaca (Other)
Responsible Party: Principal Investigator, Sabina López Toledo, Professor Investigator, Universidad Autónoma Benito Juárez de Oaxaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-04/2023
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: DIABETES Mellitus Type 2 Not Well Controlled
Keywords: DIABETES MELLITUS; Functional foods; metformin; biochemical markers; flax
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with flaxseed (Experimental): Participants in the intervention group will be given 16 g of ground flaxseed per day for 3 months.
  Interventions: Dietary Supplement: flaxseed
- Control group (No Intervention): control group, without intervention.

INTERVENTIONS:
Dietary Supplement: flaxseed — Participants in the intervention group will be given 16 g of ground flaxseed per day for 3 months.
  Arms: Intervention with flaxseed

SUMMARY:
Type 2 Diabetes Mellitus represents one of the most important health emergencies of this century Although it is known that insulin resistance is reversible and that type 2 diabetes mellitus is controllable with a change towards a healthy lifestyle, the population ignores these recommendations and continues with their unhealthy habits. Thus, the number of patients continues to grow exponentially, which leads to an increase in economic expenditure on health. This is why non-pharmacological measures are sought that favor the reduction of glycemia in patients with Diabetes Mellitus where the consumption of functional foods is a good alternative for the treatment of this chronic disease. Flaxseed is a food characterized by its nutritional properties, highlighting its content of alpha linoleic acid, flax lignans, and secoisolariciresinol diglucosides. The latter have antioxidant, lipid-lowering and hypoglycemic effects, which makes it an excellent option as a functional treatment for type 2 diabetes.

The aim of this study is to assess the adjuvant effects of flaxseed consumption (14 gr of flaxseed) on biochemical markers (glucose, glycosylated hemoglobin, total cholesterol, triglycerides, LDL cholesterol and HDL cholesterol) in adult patients (30 to 70 years) with type 2 diabetes mellitus in Oaxaca.

Procedures Patients who sign the informed consent will be assigned a group according to the following: if they have an even number in their file, they will be part of the control group (A), and if they have an odd number, they will be part of the intervention group B.

Group A. They will be given a verbal instruction to continue with the treatment established by the treating physician, and they will be given nutritional guidance with the help of the healthy eating plate.

Group B. They will be given verbal instructions to continue with the treatment established by the treating physician, they will be given nutritional guidance with the help of the healthy eating plate and they will be given a leaflet with written instructions and photos on how to consume flaxseed and its benefits.

The researchers will purchase, package and provide the flaxseed powder to the members of group B. The flaxseed will be delivered in packages with 16 gr of ground flaxseed each, which will be given to the patients for daily consumption.

DETAILED DESCRIPTION:
Researchers Dra. Sabina López Toledo (Responsible) Maria Cruz Pineda De la Cruz General objective To assess the adjuvant effects of flaxseed consumption (14 gr of flaxseed) on biochemical markers (glucose, glycosylated hemoglobin, total cholesterol, triglycerides, LDL cholesterol and HDL cholesterol) in adult patients (30 to 70 years) with type 2 diabetes mellitus, who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca.

Specific objectives

1. To describe the sociodemographic variables (age, sex, occupation, marital status) of adult patients (30 to 70 years) with type 2 diabetes, who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca.
2. Describe the clinical characteristics (time of disease evolution, type of treatment, control and comorbidities) of adult patients (30 to 70 years) with type 2 diabetes who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca.
3. Assess the biochemical parameters (glucose, glycosylated hemoglobin, total cholesterol, triglycerides, LDL cholesterol and HDL cholesterol) of adult patients (30 to 70 years) with type 2 diabetes who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca, prior to consuming flaxseed and three months after regular consumption of flaxseed.
4. Apply a nutritional intervention to two groups: Group A) Teaching about the healthy eating plate and Group B) Teaching about the healthy eating plate and indicating the consumption of flaxseed.
5. To evaluate the effect of flaxseed consumption on biochemical markers (glucose, glycosylated hemoglobin, total cholesterol, triglycerides, LDL cholesterol and HDL cholesterol of adult patients (30 to 70 years) suffering from type 2 diabetes, who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca.
6. To analyze the most effective possible combinations (pharmacological + non-pharmacological) for the treatment of adult patients (30 to 70 years) suffering from type 2 diabetes, who attend the Nutrition outpatient clinic of the Regional Hospital in Oaxaca.

Justification Type 2 Diabetes Mellitus represents one of the most important health emergencies of this century. It is estimated that in 2019 there were already 463 million people with diabetes mellitus worldwide and that this figure may increase to 578 million by 2030 and 700 million by 2030. million by 2045. A state of hyperglycemia is associated with acute and chronic complications, in both cases affecting the cardiovascular system, mainly the blood vessels and consequently the entire body, but mainly the eyes, kidneys, arteriovenous systems and peripheral nerves. Although it is known that insulin resistance is reversible and that type 2 diabetes mellitus is controllable with a change towards a healthy lifestyle, the population ignores these recommendations and continues with their unhealthy habits. Thus, the number of patients continues to grow exponentially, which leads to an increase in economic expenditure on health. This is why non-pharmacological measures are sought that favor the reduction of glycemia in patients with Diabetes Mellitus where the consumption of functional foods is a good alternative for the treatment of this chronic disease. Flaxseed is a food characterized by its nutritional properties, highlighting its content of alpha linoleic acid, flax lignans, and secoisolariciresinol diglucosides. The latter have antioxidant, lipid-lowering and hypoglycemic effects, which makes it an excellent option as a functional treatment for type 2 diabetes.

Description of the procedures Patients who sign the informed consent will be assigned a group according to the following: if they have an even number in their file, they will be part of the control group (A), and if they have an odd number, they will be part of the intervention group B.

Group A. They will be given a verbal instruction to continue with the treatment established by the treating physician, and they will be given nutritional guidance with the help of the healthy eating plate.

Group B. They will be given verbal instructions to continue with the treatment established by the treating physician, they will be given nutritional guidance with the help of the healthy eating plate and they will be given a leaflet with written instructions and photos on how to consume flaxseed and its benefits.

Phase 3. Flaxseed administration The researchers will purchase, package and provide the flaxseed powder to the members of group B. The flaxseed will be delivered in packages with 16 gr of ground flaxseed each, which will be given to the patients for daily consumption (one 8 gr spoonful of flaxseed in the morning snack and one 10 gr spoonful of flaxseed in the morning snack).

ELIGIBILITY:
Inclusion Criteria:

* Oaxaca individuals between 30 and 70 years old.
* patients who attended the Nutrition outpatient clinic at the Oaxaca Hospital President "Benito Juárez" diagnosed at most one year ago and who agreed to participate in the study by signing the informed consent.
* Patients with a diagnosis of uncontrolled type 2 diabetes, evidenced by biochemical markers, with a maximum validity of 1 month (fasting blood glucose greater than 140 and glycosylated hemoglobin greater than 6.5%).
* Patients with regular attendance at the outpatient clinic, for at least 3 consecutive months.

Exclusion Criteria:

* Patients diagnosed with chronic kidney disease on renal function replacement therapy.
* Patients with glucose disorders secondary to autoimmune diabetes, thyroid diseases or insulin-producing tumors.
* Patients with a medical history of poor drug adherence.
* Patients with adequate glycemic control evidenced by clinical laboratory tests for at least 2 months.
* Patients who do not have a means of contact for follow-up.
* Patients who are pregnant and have gestational diabetes.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose concentration | Base and through study completion, an average of 12 weeks
  Normal 70 - 99 mg/ dl Prediabetes 100 - 125 mg/ dl Diabetes >126 mg/dl
Glycosylated hemoglobin concentration | Base and through study completion, an average of 12 weeks
  Normal <5.6% Prediabetes 5.7 % - 6.4 % Diabetes >6.5%
Total cholesterol concentration | Base and through study completion, an average of 12 weeks
  Normal values should be less than 200 mg/dl
Triglycerides concentration | Base and through study completion, an average of 12 weeks
  Normal values should be less than 150 milligrams per deciliter (mg/dl) in adults

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Lopez Toledo, Doctorate, Principal Investigator — Universidad Autónoma Benito Juárez de Oaxaca (UABJO)
Locations (1):
- Hospital Regional Presidente Juárez, Oaxaca City, Oaxaca, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The plan to make the study available is to publish scientific articles in journals with high scientific rigor. The data will also be uploaded to Mexico's national data repository. A data dictionary (a description of the variables, or types of data, collected for each individual) will be provided so that the data can be fully interpreted.
  The main researcher will also have the information stored in his laboratory for one year. Researchers who want the information may request it by email
Supporting Information: Study Protocol, ICF, CSR
Time Frame: supporting information will be available (March 2025) and for 1 year (March 2026).
Access Criteria: The main researcher will have the information stored in his laboratory for one year. Researchers who want the information may request it

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT06683235/Prot_ICF_000.pdf